CLINICAL TRIAL: NCT07164183
Title: Prospective, Multicenter, Open-label, Randomized, Parallel Groups Clinical Study to Compare Efficacy and Safety of Indinol Forto® 200 mg Capsules (LLC Alcea, Russia) and Visanne 2 mg Tablets (BAYER AG, Germany) in Treatment of Endometriosis
Brief Title: Clinical Study to Compare Efficacy and Safety of Indinol Forto® 200 mg Capsules and Visanne 2 mg Tablets in Treatment of Endometriosis
Acronym: Baikal
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alcea (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND-III-2024
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: Endometriosis; Pelvic pain; Indinol Forto; indole-3-carbinol
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — indole-3-carbinol; dienogest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Participants receive Indinol Forto 200 mg capsules orally twice a day during 24 weeks
  Interventions: Drug: Indole-3-carbinol
- Arm 2 (Active Comparator): Participants receive Visanne 2 mg tablets orally once a day during 24 weeks
  Interventions: Drug: Dienogest

INTERVENTIONS:
Drug: Indole-3-carbinol — Indinol Forto (indolecarbinol (indole-3-carbinol)) 200 mg capsules orally twice a day during 24 weeks
  Arms: Arm 1
Drug: Dienogest — Visanne (dienogest) 2 mg tablets orally once a day during 24 weeks
  Arms: Arm 2

SUMMARY:
Prospective open-label randomized parallel groups study to compare efficacy and safety of Indinol Forto® 200 mg capsules and Visanne 2 mg tablets in treatment of endometriosis. This is phase 3 study, based on hypothesis of non-inferiority.

DETAILED DESCRIPTION:
Prospective open-label randomized parallel groups study to compare efficacy and safety of Indinol Forto® 200 mg capsules and Visanne 2 mg tablets in treatment of endometriosis. This is phase 3 study, based on hypothesis of non-inferiority.

The study population consists of females from 18 to 45 years old inclusively at the moment of screening who have been surgically (laparoscopy or laparotomy) diagnosed with endometriosis within not more than 60 months and not less than 2 weeks of study entry, and reported at least moderate pelvic pain within minimum 2 months of study entry.

Study participants are observed during 1 menstrual cycle during screening period (Screening Cycle). Participants who meet inclusion criteria and don't meet exclusion criteria will be randomly assigned to one of two treatment arms (Group 1: Indinol Forto® 200 mg capsules two times per day or Group 2: Visanne 2 mg tablets once per day). After observation on treatment during 24 weeks (monthly Visits 1-7) the study subjects enter post-treatment period and are observed for one more month (Post-Treatment Period, Visit 8).

Visual Analog Scale (VAS) is used in the study as the main tool for assessment of daily pelvic pain. Cyclic and non-cyclic pain, as well as intensity of vaginal bleeding are assessed daily during the study.

The study primary efficacy endpoint is the change in average daily pelvic pain score (cyclic and non-cyclic, combined) during the 6th treatment period (interval between Visit 6 and Visit 7) in comparison to the Screening period.

ELIGIBILITY:
Inclusion Criteria:

1. The participant provides written informed consent for participation in the study in accordance with current legislation.
2. Female participants in reproductive/premenopausal period from 18 to 45 years old inclusively (at the moment of signing informed consent).
3. Participants have been surgically (laparoscopy or laparotomy) diagnosed with endometriosis (ICD code #80) within not more than 60 months and not less than 2 weeks of study entry, stage I-III according to endometriosis revised classification of American Fertility Society (R-AFS, 1985)).
4. Participant has had spontaneous, (i.e., without hormonal therapy) regular, menstrual cycles with a cycle length between 24 to 38 days (inclusive) for the past 2 cycles before Visit 0 and during screening period.
5. Participant has no current indications for surgical treatment of endometriosis.
6. Participant has had endometriosis-related pelvic pain assessed with visual analogue scale (VAS) and defined as average daily pain score ≥3.5 cm during 2 menstrual cycles prior to screening (assessed by the participant retrospectively at the moment of screening) and during screening menstrual cycle (according to the data from the participant's diary completed daily).
7. Presence of other symptoms of endometriosis (e.g. dysmenorrhea, dyspareunia, dyschezia, data of ultrasound imaging, or magnetic resonance imaging (MRI).
8. The participant agrees to use highly effective contraception methods described in the protocol from the time of signing informed consent through the whole duration of the study and for 2 months after the study completion.
9. Negative pregnancy test.
10. Participant completed daily diary on minimum 75% of days during screening menstrual cycle.

Exclusion Criteria:

1. Presence of contraindications to Indinol Forto (indolcarbinol)
2. Presence of contraindications to Visanne (dienogest)
3. Participant had undiagnosed (unexplained), abnormal, vaginal or urinary tract bleeding within the past 6 months before screening (Visit 0).
4. Participant has chronic pelvic pain not caused by endometriosis, but other gynecological or urological disorders (consequences of inflammatory process, uterine fibroids, pelvic congestion syndrome, etc.).
5. Participant has chronic, non-pelvic pain not caused by endometriosis that requires chronic analgesic or other chronic therapy (including, but not limited to, fibromyalgia, chronic back pain or chronic headaches).
6. Endometrioid cysts ≥ 3 cm.
7. Participant has a surgical history of hysterectomy and/or bilateral oophorectomy; premature ovarian failure. Note: Participants who have undergone surgical sterilization (eg, bilateral salpingectomy, tubal ligation) are permitted in the trial.
8. Participant has a clinically significant gynecologic condition identified in the screening evaluation including, but not limited to, ovarian cysts larger than 3 cm and present longer than 4 months, an active sexually transmitted disease, etc. Note: Participants may be rescreened after completing treatment for infection or for simple ovarian cysts.
9. Participant with endometriosis-related pelvic pain who didn't respond to previous treatment with combined oral contraceptives, GnRH agonists or antagonist, progestins or aromatase inhibitors. Note: Participants who demonstrated partial response or interrupted their treatment due to side effects, may be enrolled in the study.
10. History of malignancy, including suspected malignization of endometriomas within ≤5 years before signing informed consent, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
11. Severe renal failure (glomerular filtration rate calculated with Cockcroft-Gault formula is below 30 ml/min/1,73 m2).
12. Systolic blood pressure >160 mm Hg or diastolic blood pressure >90 mm Hg during screening period.
13. Clinically significantly abnormal laboratory tests at Screening, including: alkaline phosphatase (AP), alanine aminotransferase (ALT, SGPT), aspartate aminotransferase (AST, SGOT) >200% of the upper limit of normal, or total bilirubin >150% of the upper limit of normal; hemoglobin <10 g/dl, white blood cell count <2500 in mm³, neutrophil count <1500 in mm³, platelet count <100 х 10³/mm³.
14. Hyperthyroidism (TSH below 0.4 mU/L) or hypothyroidism (TSH above 4.0 mU/L).
15. Positive pregnancy test (including pregnancy within 3 months prior to screening) or lactation period.
16. Other medical conditions that, in the judgment of the Investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results.
17. History of alcohol or substance abuse.
18. Participation in a clinical study within 90 days before screening.
19. Other reasons that, in the judgment of the Investigator, may interfere with participation in the study or may lead to unreasonable risks.
20. Conditions requiring surgery in the period of the study.
21. Conditions requiring therapy prohibited by the study protocol.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female participants in reproductive/premenopausal period from 18 to 45 years old inclusively (at the moment of signing informed consent).
Enrollment: 290 (Estimated)
Dates: Start 2025-09-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Average daily pelvic pain score, combined | Visit 7 (week 24)
  Change in average daily VAS (in mm) endometriosis-related pelvic pain score (cyclic and non-cyclic, combined) during Treatment Period 6 (assessed at Visit 7) in comparison to Screening Cycle as reported in the participant's diary.

SECONDARY OUTCOMES:
Average daily pelvic pain score, cyclic | Visit 7 (week 24)
  Change in average daily VAS (in mm) endometriosis-related pelvic pain score (cyclic) during Treatment Periods in comparison to Screening Cycle as reported in the participant's diary.
Average daily pelvic pain score, non-cyclic | Visit 7 (week 24)
  Change in average daily VAS (mm) endometriosis-related pelvic pain score (non-cyclic) during Treatment Periods in comparison to Screening Cycle as reported in the participant's diary.
Proportion of participants with improvement | Visit 7 (week 24)
  Proportion of participants with more than 10 mm reduction (at least minimal clinically significant change) in average daily pelvic pain score (cyclic, non-cyclic and combined) during Treatment Period 6 (assessed at Visit 7) in comparison to Screening Cycle
Change in signs and symptoms of endometriosis assessed in B&B scale | Visit 8 (week 28)
  Change in signs and symptoms of endometriosis (including dyspareunia), assessed with B&B scale at visits 2, 4, 7, 8 in comparison to baseline (Visit 1).
Proportion of participants with full recovery | Visit 7 (week 24)
  Proportion of participants with complete absence of endometriosis symptoms, assessed with B&B scale at Visit 7.
Proportion of participants with recurrence of endometriosis | Visit 8 (week 28)
  Proportion of participants with recurrence of endometriosis symptoms, assessed with B&B scale at Visit 8.
Quality of life change | Visit 8 (week 28)
  Change in the quality of life assessment at Visits 2-8 in comparison to Visit 1 according to the EPH-30 questionnaire (total and in each of the modules).
Menstruation duration | Visit 8 (week 28)
  Change in average duration of menstruation (in days) during Treatment Period and In Post-Treatment Period in comparison with Screening Cycle.
Menstruation intensity | Visit 8 (week 28)
  Proportion of participants with more intensive, less intensive and normal menstruation during Treatment Period and In Post-Treatment Period in comparison with Screening Cycle.
Irregular vaginal bleeding | Visit 8 (week 28)
  Proportion of participants with irregular vaginal bleeding during Treatment Periods and in Post-Treatment Period in comparison with Screening Cycle.
Proportion of participants with amenorrhea | Visit 8 (week 28)
  Proportion of participants with amenorrhea during Treatment Periods and in Post-Treatment Period.
Number of menstruations | Visit 8 (week 28)
  Number of menstruations (counted on day 1) registered during Treatment Periods.
Menstrual Cycle Duration | Visit 7 (week 24)
  Duration of the last menstrual cycle (from day 1 of the previous menstruation to day 1 of the last menstruation) registered in the period from Visit 4 to Visit 7 (if applicable).
Endometriosis lesions size | Visit 7 (week 24)
  Change in size of the biggest ovarian endometriosis lesion at Visit 7 in comparison to Screening ultrasound assessment.

OTHER OUTCOMES:
Estrogens level | Visit 7 (week 24)
  Proportion of subjects with minimum 5% decrease of estrogens (estrone and estradiol) level.
Estrogens index | Visit 7 (week 24)
  Proportion of subjects with minimum 5% increase of estrogens (estrone/estradiol) metabolic index.
Ferritin level | Visit 7 (week 24)
  Proportion of subjects with ferritin below 20 ng/ml at Visit 0 and at Visit 7.

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Rostov-on-Don
  - Research Site, Ryazan
  - Research Site, Saint Petersburg
  - Research Site, Smolensk
  - Research Site, Tver'
  - Research Site, Yaroslavl